CLINICAL TRIAL: NCT03475680
Title: Mechanical Bowel Preparation and Oral Antibiotics Before Colon Cancer Surgery: a Multi Center Double-Blinded Randomized Controlled Trial (COLONPREP Study)
Brief Title: Mechanical Bowel Preparation and Oral Antibiotics Before Colon Cancer Surgery
Acronym: COLONPREP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of inclusions
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P161202J
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer
Keywords: Mechanical Bowel Preparation (MBP); Oral antibiotics; Colon cancer surgery; Surgical site infection
MeSH Terms: conditions — Colonic Neoplasms; Surgical Wound Infection | interventions — Gentamicins; Ornidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind : both participants and investigators are unaware of the intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1) " MBP and oral antibiotics " group (Experimental): Sennosides colonic preparation Oral Gentamycin Oral Ornidazole
  * Sennosides colonic preparation (X-PREP) :
    1 per day, on day -2 and day -1.
  * Gentamycin :
    80 mg, 4 per day, on day -2 and day -1; Liquid forms in individual vials.
  * Ornidazole :
    1. g per day (2 tablet per day), on day -2 and day -1; In tablets.
  Interventions: Drug: Sennosides colonic preparation; Drug: Oral Gentamycin; Drug: Oral Ornidazole
- 2) " MBP alone " group (Placebo Comparator): Sennosides colonic preparation Oral placebo Gentamycin Oral placebo Ornidazole
  * Sennosides colonic preparation (X-PREP) :
    1 per day, on day -2 and day -1.
  * Placebo for oral gentamycin:
  Same presentation as oral gentamycin x4 per day on day -2 and day -1. - Placebo for oral ornidazole : Same presentation as oral ornidazole
  1g per day (2 tablet per day) on day -2 and day -1.
  Interventions: Drug: Sennosides colonic preparation; Drug: Oral placebo Gentamycin; Drug: Oral placebo Ornidazole
- 3) " Oral antibiotics alone " group (Experimental): Oral Gentamycin Oral Ornidazole
  * Gentamycin :
    80 mg, 4 per day, on day -2 and day -1; Liquid forms in individual vials.
  * Ornidazole :
    1. g per day (2 tablet per day), on day -2 and day -1; In tablets.
  Interventions: Drug: Oral Gentamycin; Drug: Oral Ornidazole
- 4) " No preparation " group (Placebo Comparator): Oral placebo Gentamycin Oral placebo Ornidazole
  - Placebo for oral gentamycin : Same presentation as oral gentamycin x4 per day on day -2 and day -1
  - Placebo for oral ornidazole : Same presentation as oral ornidazole
  1g per day (2 tablet per day) on day -2 and day -1
  Interventions: Drug: Oral placebo Gentamycin; Drug: Oral placebo Ornidazole

INTERVENTIONS:
Drug: Sennosides colonic preparation — Mechanical bowel preparation :
  Sennosides colonic preparation (X-PREP)
  1 per day, on day -2 and day -1
  Arms: 1) " MBP and oral antibiotics " group; 2) " MBP alone " group
Drug: Oral Gentamycin — Gentamycin 80 mg, 4 per day, on day -2 and day -1; Liquid forms in individual vials
  Arms: 1) " MBP and oral antibiotics " group; 3) " Oral antibiotics alone " group
Drug: Oral Ornidazole — Oral Ornidazole :
  Ornidazole
  1 g per day (2 tablet per day), on day -2 and day -1; In tablets
  Arms: 1) " MBP and oral antibiotics " group; 3) " Oral antibiotics alone " group
Drug: Oral placebo Gentamycin — Placebo for oral gentamycin :
  Same presentation as oral gentamycin x4 per day on day -2 and day -1
  Arms: 2) " MBP alone " group; 4) " No preparation " group
Drug: Oral placebo Ornidazole — Placebo for oral Ornidazole :
  Same presentation as oral ornidazole
  1g per day (2 tablet per day) on day -2 and day -1
  Arms: 2) " MBP alone " group; 4) " No preparation " group

SUMMARY:
This study aims to demonstrate that a preoperative combination of mechanical bowel preparation and oral antibiotics, before elective laparoscopic colon cancer surgery, is associated with a reduction of postoperative surgical site infection rate, as compared to mechanical bowel preparation alone, oral antibiotics alone, or no colonic preparation.

Our Hypothesis is that a preoperative colonic preparation including a combination of mechanical bowel preparation and oral antibiotics before elective laparoscopic colon cancer surgery is associated with a reduced rate of 30-day postoperative surgical site infection, as compared to mechanical bowel preparation alone, oral antibiotics alone, or no colonic preparation.

DETAILED DESCRIPTION:
Preoperative mechanical bowel preparation (MBP) has been proposed in an attempt to reduce the colonic fecal load and to limit the risk of surgical site contamination, thus theoretically limiting the risk of postoperative SSI. However, several randomized-controlled trials (RCT) and meta-analyses, have suggested the absence of benefit, in term of postoperative morbidity, of preoperative MBP before elective colon cancer surgery. A meta-analysis of RCT, comparing MBP to no-MBP before elective colon cancer surgery, even suggested that MBP could be associated with an increased SSI rate, as compared to no-MBP. These results led the latest French surgical guidelines of the Société Française de Chirurgie Digestive (SFCD) to recommend the absence of MBP before elective colon cancer surgery.

However, recent studies suggested that the adjunction of oral antibiotics during MBP could help efficiently reduce the risk of postoperative SSI. Indeed, a recent meta-analysis of RCT have suggested that patients preoperatively receiving both MBP and oral antibiotics were exposed to a significantly reduced risk of postoperative SSI, as compared to patients receiving only preoperative MBP. This result was confirmed in a recent RCT which compared preoperative MBP and oral antibiotics versus MBP alone in a heterogeneous population of patients who underwent laparoscopic colonic or rectal surgery. This latter study reported a 50% reduction of SSI rate in the "MBP and oral antibiotics" group, as compared to the "MBP alone" group. Finally, three recent large retrospective registry studies compared the outcomes of four different strategies of preoperative colonic preparation before colorectal surgery: 1) MBP and oral antibiotics, 2) MBP alone, 3) Oral antibiotics alone, and 4) No colonic preparation. However, to date, no RCT has compared the "No preparation" group, which is the gold standard according to the international and French guidelines, to the "MBP and oral antibiotics" group.

The present study is therefore the first double-blinded RCT to compare the SSI rate for 4 types of colonic preparation before elective laparoscopic colonic surgery: 1) MBP and oral antibiotics, 2) MBP alone, 3) Oral antibiotics alone, and 4) No preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or more
* Scheduled to undergo elective restorative laparoscopic segmental colectomy for colon cancer
* With Signed consent
* And affiliated to the French social security system

Exclusion Criteria:

* Emergent surgery
* Scheduled total or subtotal colectomy (defined as a colectomy extended from the right colon to a least the left colonic angle)
* Scheduled transverse colectomy
* Scheduled associated proctectomy
* Scheduled associated concomitant resection of another organ (liver, etc.), except the abdominal wall
* Previous segmental colectomy
* Associated inflammatory bowel disease
* Active bacterial infection at the time of surgery or recent antimicrobial therapy (up to 2 weeks before surgery)
* Patients with known colonization with multidrug-resistant enterobacteriacea
* History of allergy or contraindication to the Ornidazole, Gentamycin, X-PREP or to any of the excipients of the drugs used.
* Cirrhosis of grade B and C (Child-Pugh classification)
* Myasthenia
* Allergy to one of the other treatments administered for the purpose of the trial (including betadine)
* Patient suffering from severe central neurologic diseases, fixed or progressive.
* Pregnant patients
* Refusal to participate or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Postoperative 30-day surgical site infection (SSI). | 30 days
  SSI will be defined and classified as superficial, deep and/or organ-space infection on the basis of validated and well-defined criteria developed by the Centers for Disease Control and Prevention (CDC), validated in French by the Comité technique des infections nosocomiales et des infections liées aux soins

SECONDARY OUTCOMES:
Overall postoperative morbidity | 30 days
  Including all postoperative complications occurring within 30 days after surgery, defined and classified according to the Clavien-Dindo classification.
Severe postoperative morbidity | 30 days
  Including all complications graded 3 or more according to the Clavien-Dindo classification, and occurring within 30 days after surgery.
Postoperative mortality | 30 days
  Including all deaths occurring within 30 days after surgery.
Postoperative anastomotic leakage | 90 days
  Defined as the passing of any intra-colonic content (air, liquid, intestinal content, or radiological contrast) through an anastomosis or by an peri-anastomotic abscess, even in the absence of intra-colonic content leak through the anastomosis, observed in drainages, surgical incision, vagina, during a surgical procedure or on a radiological examination, occurring within 90 days after surgery.
Postoperative length of hospital stay | Day of hospital discharge
  Calculated from the day of surgery to the day of hospital discharge.
Unplanned hospitalization | 90 days
  Defined as any unplanned hospitalization between surgery and postoperative day 90.
Tolerance of the colonic preparation | The day before surgery
  Evaluated using a dedicated tolerance of the colonic preparation questionnaire performed the evening before surgery.
Clostridium difficile colitis occurrence | 30 days
  Defined as clinical symptoms of clostridium difficile colitis with at least 1 stool sample positive for Clostridium difficile toxin A/B as detected by enzyme-linked immunosorbent assay within 30 days after surgery.
Rate of multi-resistant bacteria carriage | The day before or the day of surgery
  Defined as rate of multi-resistant bacteria carriage
Date of adjuvant chemotherapy beginning | During 90 days
  If indicated

CONTACTS AND LOCATIONS:
Locations (1):
- Service de chirurgie Colorectale / Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available